CLINICAL TRIAL: NCT02923557
Title: Prophylactic Intravesical Chemotherapy to Prevent Bladder Recurrence After Nephroureterectomy for Primary Upper Tract Urothelial Carcinoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xuesong Li, Associated Professor, Peking University First Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IUPU-16-UTUC-2
Record Dates: First submitted 2016-10-01; First posted 2016-10-04 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Bladder Recurrence; Upper Tract Urothelial Carcinoma; Nephroureterectomy
MeSH Terms: interventions — pirarubicin

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Blank control (No Intervention): do not use prophylactic intravesical chemotherapy.
- Single intravesical instillation (Experimental): intravesical instillation within 24 hours postoperatively
  Interventions: Drug: Pirarubicin

INTERVENTIONS:
Drug: Pirarubicin — single immediate intravesical dose of pirarubicin (THP) intravesical therapy (THP 40 mg for 30 min) within 24 hours of nephroureterectomy.
  Arms: Single intravesical instillation

SUMMARY:
This clinical trial is designed to evaluate the efficacy of single immediate intravesical chemotherapy instillation in the prevention of bladder recurrence after nephroureterectomy for primary upper tract urothelial carcinoma (UTUC) patients.

DETAILED DESCRIPTION:
INTRODUCTION

Upper tract urothelial carcinomas (UTUC) are relatively uncommon compared to bladder cancer and account for only 5-10% of urothelial carcinomas, with an estimated annual incidence in Western countries of ~2 cases per 100,000 inhabitants. In 17% of cases, concurrent bladder cancer is present. Recurrence in the bladder after management of UTUC occurs in 22-47% of UTUC patients, compared with 2-6% in the contralateral upper tract. At our institution, we reported that 30.8% of UTUC patients developed intravesical recurrence, which was in line with the global trend.

Generally speaking, the field cancerization hypothesis and intraluminal seeding are currently the two main concepts to explain multifocality of urothelial cancer and the recurrent bladder tumor. Independent multiclonal tumor development after carcinogenic exposure of the entire urothelial and intraluminal implantation followed by clonally induced single progenitor cell evolution are the mechanisms suggested. While the two mechanisms could co-exist, the intraluminal seeding hypothesis is becoming more prevalent with the emergence of more evidence from molecular studies. Thus postoperative intravesical chemotherapy could potentially remove the implantation cell and prevent recurrence. While intravesical instillation is widely used to prevent recurrence after transurethral resection for primary bladder tumors, there is still no consensus on the prophylactic capability of intravesical chemotherapy in preventing bladder recurrence after nephroureterctomy for UTUC. According to a previous prospective, multicentre, randomised clinical trial, a single postoperative dose of intravesical mitomycin C appears to reduce the risk of a bladder tumour within the first year following nephroureterectomy for UTUCs.

AIM OF THE WORK This clinical trial is designed to evaluate the efficacy of single immediate intravesical chemotherapy instillation in the prevention of bladder recurrence after nephroureterectomy for UTUCs.

ELIGIBILITY:
Inclusion Criteria:

* Suspected UTUC patients without history of bladder tumor.
* Suspected UTUC patients without synchronous bladder tumor.
* Suspected UTUC patients without contralateral UTUCs.

Exclusion Criteria:

* Patients with history of bladder tumor.
* Patients with synchronous bladder tumor.
* Patients with contralateral UTUCs.
* Patients with advanced stage (T4).
* Patients with other malignant tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
intravesical recurrence-free survival | three years after surgery

SECONDARY OUTCOMES:
cancer-specific survival | three years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Frist Hospital, Beijing, Beijing Municipality, China